CLINICAL TRIAL: NCT00514553
Title: Deliberation With and Without Attention: Can We Enhance Informed Choices About Invasive Prenatal Testing? A Proof of Principle Study
Brief Title: Informed Choice Regarding Invasive Prenatal Testing
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 070204; 07-HG-0204
Record Dates: First submitted 2007-08-09; First posted 2007-08-10 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-05-31

CONDITIONS: Pregnancy - Prenatal Testing
Keywords: Prenatal Testing; Test Decision-Making; Decision-Making Intervention; Theory of Unconscious Thought; Informed Choice; Decision Making; Counseling

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This study will compare the effectiveness of two interventions to help women make informed choices about whether or not to undergo an invasive procedure (amniocentesis or chorionic villus sampling) for prenatal testing. The interventions are: 1) conscious deliberation (getting women to focus on and engage in the decision) and 2) unconscious deliberation (getting women not to focus on the decision). Studies suggest that some women are ambivalent about their decisions regarding invasive prenatal testing and those with the most ambivalence experience greater conflict about the decision. Techniques to reduce ambivalence through conscious or unconscious deliberation might lead to better informed choices. The two methods will also be compared with standard counseling for prenatal testing decisions.

Women 18 years of age or older who are referred for prenatal genetic counseling to consider invasive prenatal testing and who have not previously undergone prenatal testing may be eligible for this study.

Participants complete a questionnaire before and after receiving standard genetic counseling. They are then randomly assigned to one of three study groups:

* Standard genetic counseling (control group): Receives no further intervention beyond standard counseling.
* Conscious deliberation: Participants complete a form that focuses their attention on the pros and cons of invasive prenatal testing. This is followed by a brief questionnaire to evaluate time spent thinking about the session and the ease of completing the session.
* Unconscious deliberation: Participants are provided a distraction task to complete during the session, such as a word or number puzzle and are told they will be asked about their decision regarding invasive prenatal testing at the end of the session. This is followed by a brief questionnaire to evaluate time spent thinking about the session and the ease of completing the session.

Participants are contacted by telephone 1 month after the counseling session to find out what they decided regarding invasive prenatal testing and to assess any conflict they experienced about the decision.

...

DETAILED DESCRIPTION:
This study will compare the efficacy of two interventions aimed at facilitating informed choice about invasive prenatal testing: a) deliberation with attention and b) deliberation without attention. Deliberation with attention is conscious engagement and deliberation without attention is aimed at facilitating unconscious engagement. These will be compared with standard counseling for prenatal testing decisions. As a proof of principle study, the overall study goal is to demonstrate that the interventions have the desired effect on the variables hypothesized to be proximal to the primary endpoint. In this case, we aim to demonstrate an effect for both interventions on the outcome of value-behavior consistency and to determine effect sizes for estimating the sample size needed for a clinical trial.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Women referred for prenatal genetic counseling to consider invasive prenatal testing who have not previously undergone prenatal testing.
* Women who are ambivalent about undergoing prenatal testing. They will be screened for ambivalence by answering no to a question about whether they have decided to undergo prenatal testing and yes to a close-ended question about whether you have mixed or conflicting feelings toward undergoing testing.
* Women must be greater than or equal to 18 years old.
* Participants must speak English
* Participants must be competent to consent to participate in the study.

EXCLUSION CRITERIA:

* Men
* Participants less than 18 years of age.
* Participants who cannot speak English.
* Participants who are not competent to consent to participate in the study.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2007-08-07; Study Completion 2011-05-31

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] O'Connor AM, Jacobsen MJ, Stacey D. An evidence-based approach to managing women's decisional conflict. J Obstet Gynecol Neonatal Nurs. 2002 Sep-Oct;31(5):570-81. doi: 10.1111/j.1552-6909.2002.tb00083.x. PMID 12353737
- [Background] Bekker HL, Hewison J, Thornton JG. Understanding why decision aids work: linking process with outcome. Patient Educ Couns. 2003 Jul;50(3):323-9. doi: 10.1016/s0738-3991(03)00056-9. PMID 12900106
- [Background] Wilson TD, Schooler JW. Thinking too much: introspection can reduce the quality of preferences and decisions. J Pers Soc Psychol. 1991 Feb;60(2):181-92. doi: 10.1037//0022-3514.60.2.181. PMID 2016668